CLINICAL TRIAL: NCT00334009
Title: Impact of Catecholamine-O-Methyl-Transferase Enzyme Activity on Clinical and Biological Parameters in Patients After Cardiac Surgery.
Brief Title: Catecholamine-O-Methyl-Transferase(COMT)-Polymorphism in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Austin Health (Other Government)
Other Study IDs: H2005/02320
Record Dates: First submitted 2006-06-05; First posted 2006-06-06 (Estimated); Last update posted 2008-03-06 (Estimated); Status verified 2008-03

CONDITIONS: Cardiac Surgery
Keywords: Cardiac Surgery; Cardiopulmonary Bypass; COMT-Polymorphism; Vasoplegia; Catecholamines; Acute Renal Failure
MeSH Terms: conditions — Vasoplegia; Acute Kidney Injury

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Although clinical risk factors for postoperative development of vasodilatory shock and acute renal failure have been identified; there is a considerable proportion of patients undergoing cardiac surgery where this syndrome cannot be predicted.

We sought to investigate the impact of Catecholamine-O-Methyltransferase (COMT) polymorphism on the duration of vasodilatory shock and other important clinical outcomes in cardiac surgery patients.

COMT is a key enzyme in the degradation of catechols eg. catecholamines. 25% of the population have a low activity (L/L) of this enzyme. Sustained low COMT activity is associated with an altered metabolic profile of catecholamines and their degradation products.

The process of cardiopulmonary bypass (CPB)over-activates some of the same mechanisms the body uses to defend itself against severe infection. One of the main overactive defence mechanisms is the release of highly toxic compounds derived from oxygen - a process called 'oxidative-stress'. Increased reactive oxygen species (ROS) generation can lead to inactivation of biologic mediators, including catecholamines. It is well established that some radicals autoxidizes catecholamines, including DA, NE, and epinephrine and contribute significantly to vasoplegia.

As part of this study, we will take six 2.7mL samples of blood, collected before, and after the operation, from the arterial catheter routinely inserted in every patient. This blood will be used to measure COMT genotype, the concentration of plasma-catecholamines as well as marker of oxidative stress.

Our plan is to enrol patients undergoing cardiac surgery if the use of the CPB is planned.

DETAILED DESCRIPTION:
Aim of the study

To explore if there is an impact of LL COMT genotype on clinical and biological outcome variables in patients undergoing cardiac surgery compared to HH genotype.

Background

Cardiac surgery has been shown to be an effective method for prolonging life in patients with severe coronary artery disease or valvular disease or a combination thereof.

Catechol-O-Methyl-Transferase (COMT) catalyses the O-methylation of biologically active catechols and is responsible for the degradation of catecholamines and catecholestradiols.

COMT is an intracellular enzyme, which is widely distributed throughout most of all human tissues (Roth, Maennistoe) Because COMT is expressed ubiquitously, it appears that the COMT genotype significantly affects levels of catecholamines throughout the body.

25 % of Caucasians are homozygous for low COMT activity, (COMT LL=Met/Met), 25% are homozygous for high activity of COMT (COMT HH=Val/Val), and about 50% are heterozygous (COMT HL=Val/Met). (Palmatier, Spielman, Boudikova)

Thus, COMT polymorphism may play an important role in the outcome of patients after cardiac surgery.

So far, studies due to this polymorphism exist only for chronic, non-cardiac surgery disorders like psychiatric diseases, breast cancer and alcoholism.

In a prospective observational study, we used this model of CPB-induced stress-mediated vasodilatory shock to investigate the impact of COMT polymorphism on relevant postoperative clinical outcomes. Within this model we tested the hypothesis that, in cardiac surgery patients, the LL COMT genotype is associated with alterations in catecholamine metabolism and adverse hospital outcomes such as prolonged vasopressor support and acute renal failure compared to HL and HH COMT genotype.

Patients with a L/L COMT polymorphism are probably used to higher concentrations of endogenous catecholamines, because a low COMT enzyme activity can cause an impaired degradation of catecholamines. Patients with a L/L COMT polymorphism require presumably higher catecholamines support than other patients to maintain cardiovascular stability in extreme stress-conditions occuring during CPB procedures.

Acute renal failure (ARF) is a common postoperative complication in cardiac surgery patients that is associated with increased morbidity and mortality. Catechol-O-methyltransferase (COMT) shows high activity in proximal tubular epithelial cells - target cell in ARF. We hypothesized that the COMT met158 genotype might be associated with increased risk of acute renal failure compared to COMT val158 genotype.

CPB activates components of the non-specific immune system, which leads to the generation of compounds containing oxygen free radicals. A study of 14 patients undergoing cardiac surgery found increased levels of serum lipid peroxidation products (thiobarbituric acid reactive substances) within 15 minutes of the commencement of CPB, which returned to preoperative levels by the following morning. The total serum antioxidative capacity was correspondingly decreased intraoperatively, and remained decreased at 24 hours postoperatively.

Outcomes will be the length of vasopressor support in patients with LL COMT genotype compared to patients with HL and HH COMT genotype. We hypothesize that there is a significant increase in the duration of vasopressor support in patients with LL COMT compared to patients with HL and HH COMT genotype.

Additional outcome measure and hypotheses

We hypothesize that differences similar to that seen in the duration of vasopressor support will be seen in a higher proportion of postoperative acute renal failure (increase in serum creatinine >50% from baseline to peak value), longer duration of ICU and hospital stay in LL COMT patients compared to HL and HH patients.

COMT genotype will be determined and levels of endogenous catecholamines will be measured before and after cardiac surgery. We hypothesize that higher levels of endogenous catecholamines will be measured for patients with LL COMT genotype.

Study Design - overview and rationale

COMT genotype and outcome measurements of patients after cardiac surgery will be analyzed in this study. Concentrations of plasma catecholamines and important degradation products will be determined before and after the use of CPB. The duration and dose of postoperative vasopressor support as well as stay in ICU and stay in hospital will be documented.

Data collection

age, sex, body mass index (BMI), body surface area (BSA, insulin (IDDM) or non-insulin dependent diabetes mellitus (NIDDM), arterial hypertension, hypercholesterolemia, preoperative serum creatinine, chronic obstructive pulmonary disease (COPD), smoking status, peripheral vascular disease (PVD), carotid artery disease, myocardial infarction (MI) or stroke within last six months, atrial fibrillation (AF), and grade of left ventricular dysfunction defined by the left ventricular ejection fraction using EuroScore definition. Pre-operative medication including: platelet inhibitors, ACE-inhibitors/angiotensin-II-receptor1-antagonists, beta-blocker, calcium channel blocker and statins.

Intra-operative data on type of cardiac surgery (valvular or coronary artery bypass (CABG), concomitant or complex cardiac surgery involving the ascending aorta), Redo operation, take back to operating room, electronically stored MAP and duration of CPB. The intra- and post-operative use of vasopressor (norepinephrine, epinephrine, phenylephrine, ephedrine, and metaraminol) and inotropic medications (milrinone, dobutamine)hourly until discharge from the Intensive Care Unit (ICU). We will note the lowest MAP and the lowest cardiac index (CI) every 6 hours. Postoperative serum creatinine will be measured daily. Finally, ICU and hospital length of stay as well as hospital mortality were documented.

Withdrawal The treating clinician will have the right to withdraw the patient from the study if he or she believes that continued participation is jeopardising the patient's well being.

Ethical Issues Given the potential knowledge for the future the balance of benefits and risks, we consider it ethical to proceed and seek informed consent. This is not a drug trial or an interventional trial.

Indemnity This is an investigator-initiated study and is not sponsored by industry. The investigator is a member of staff at Austin Hospital; the hospital is responsible for indemnifying the investigator in relation to this study. Warringal Private Hospital will be responsible for indemnification for patients recruited there.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective cardiac surgery (in whom CPB is planned) at the Austin Hospital and Warringal Private Hospital.

Exclusion Criteria:

* Intake of Levodopa
* Intake of COMT inhibitors (e.g. Entacapone, Tolcapone)
* Intake of monoamino oxidase inhibitors type A and B (e.g. Moclobemide, Selegiline, Rasagiline)
* Patients below 18 years of age
* oral steroids
* emergency patients (cardiac symptoms occurred < 24 hours prior to operation)
* patients receiving IV nitrates/nitroprusside sodium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 2006-06; Study Completion 2006-11

PRIMARY OUTCOMES:
duration of vasoplegia and incidence of acute renal failure following cardiopulmonary bypass

SECONDARY OUTCOMES:
length of stay in intensive care and in hospital, requirement of renal replacement therapy, mortality

CONTACTS AND LOCATIONS:
Overall Officials: Rinaldo Bellomo, MD, FRACP, Principal Investigator — Austin Health; Duska Dragun, MD, Principal Investigator — Department of Nephrology, Charite University Hospital, Berlin
Locations (1):
- Austin Hospital, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Haase-Fielitz A, Haase M, Bellomo R, Lambert G, Matalanis G, Story D, Doolan L, Buxton B, Gutteridge G, Luft FC, Schunck WH, Dragun D. Decreased catecholamine degradation associates with shock and kidney injury after cardiac surgery. J Am Soc Nephrol. 2009 Jun;20(6):1393-403. doi: 10.1681/ASN.2008080915. Epub 2009 Apr 30. PMID 19406978